CLINICAL TRIAL: NCT00797394
Title: Efficacy of Natural Extract 2007RD01 Combined With Saw Palmetto in Benign Prostatic Hyperplasia Patients Compared to Saw Palmetto
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: innoVactiv Inc. (Industry)
Responsible Party: Jocelyn Bérubé / Scientific Director, Health & Nutrition, innoVactiv inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-RD-01-CLN
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: prostate; dietary supplements; saw palmetto; canada
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Treated (Experimental)
  Interventions: Dietary Supplement: Combination of 2007RD01 and saw palmetto lipidic extract
- Control (Active Comparator)
  Interventions: Dietary Supplement: Saw palmetto lipidic extract

INTERVENTIONS:
Dietary Supplement: Combination of 2007RD01 and saw palmetto lipidic extract — Oral administration of one capsule containing a combination of 250 mg of 2007RD01 (a natural extract) and 160 mg of saw palmetto lipidic extract plus inactive fillers, twice a day between meals
  Arms: Treated
Dietary Supplement: Saw palmetto lipidic extract — Oral administration of one capsule of 160 mg of saw palmetto lipidic extract plus inactive fillers, twice a day between meals
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the combination of 2007RD01, a natural extract, and saw palmetto lipidic extract, is more effective at treating lower urinary tract symptoms associated with benign prostatic hyperplasia than saw palmetto lipidic extract alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be an adult man aged between 50 and 75
* Patient must have Benign Prostatic Hyperplasia symptoms

Exclusion Criteria:

* Patient has a malfunction of the urinary tract, is suffering from acute urinary retention, or is suffering from prostate cancer or urinary tract infection
* Patient has been subjected to surgery of the prostate, bladder or urethra
* Patient has taken a 5-alpha-reductase inhibitor in the 6-month period preceding screening
* Patient has taken an alpha-blocker in the 2-week period preceding screening

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Absolute and relative (%) change in IPSS between baseline and end of study | 90 days ±7 days

SECONDARY OUTCOMES:
Absolute and relative (%) change in IPSS between baseline and day 30 of follow-up | 30 days ±7 days
Absolute and relative (%) change in peak urinary flow between baseline and after 30 or 90 days of follow-up | 30 days ±7 days , 90 days ±7 days
Absolute and relative (%) change in post-void residual volume between baseline and after 30 or 90 days of follow-up | 30 days ±7 days , 90 days ±7 days
Change in health related quality of life between baseline and after 30 or 90 days of follow-up | 30 days ±7 days , 90 days ±7 days
Change in sexual function between baseline and after 30 or 90 days of follow-up | 30 days ±7 days , 90 days ±7 days

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Recherches Cliniques Theradev, Granby, Quebec
  - Urology South Shore Research, Greenfield Park, Quebec
  - Les Urologues Associés du CHUM, Montreal, Quebec
  - Clinique d'urologie Berger, Québec, Quebec